CLINICAL TRIAL: NCT06164197
Title: A Comparison of the Effects of Virtual Reality-Based Balance Training and Robot-Assisted Gait Training on Balance and Gait Performance in Individuals with Stroke
Brief Title: Virtual Reality Based Robotic Gait and Balance Trainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Murat Akıncı, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAGT03
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: Stroke; Virtual Reality; Lokomat; Thera-Trainer; Balance-Trainer; Robot Assisted Gait Training; Robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lokomat (Experimental)
  Interventions: Device: Lokomat; Other: Person-Specific Rehabilitation Program
- Balance Trainer (Experimental)
  Interventions: Device: Thera Trainer Balo; Other: Person-Specific Rehabilitation Program

INTERVENTIONS:
Device: Lokomat — Robot Assisted Gait Training
  Arms: Lokomat
Device: Thera Trainer Balo — Virtual Reality Based Balance Training Device
  Arms: Balance Trainer
Other: Person-Specific Rehabilitation Program — Person-Specific Rehabilitation Program

SUMMARY:
The aim of research is to examine and compare the effectiveness of virtual reality-based balance training and robot-assisted walking approaches on balance and gait in individuals post-stroke. Through the study, Investigators intend to reach conclusions regarding whether the focus should be on balance or walking training based on the Berg Balance Scale and Functional Ambulation Classification levels of stroke survivors. Subgroups will be formed in both groups based on Functional Ambulation and Berg Balance Scale scores. The balance and gait developments within these subgroups will be compared, aiming to determine at which levels balance or walking improvement is more pronounced. These findings are crucial for making the right choices in setting rehabilitation goals for individual patients.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death in adults and results in severe disability. Within the first 3 months after a stroke, 20% of patients use a wheelchair, and 70% experience walking problems. Balance problems are among the most common issues after a stroke, impacting a patient's ability to sit, stand, transfer, and walk, thereby creating a risk of falls. Additionally, balance and walking quality are vital components, with abnormalities potentially leading to abnormal walking patterns, reduced walking speed, and spatiotemporal asymmetries. Therefore, improving balance and walking is a fundamental goal in stroke rehabilitation and holds priority for many patients and their families.

Robot-assisted gait training (RAGT) is an emerging and promising technological approach in stroke rehabilitation. RAGT provides safe, high-intensity, and task-oriented walking training with ample repetitions. Repetitive tasks can enhance neuroplasticity and motor learning, resulting in improved balance and walking speed.

Robotic systems come in two types: end-effector and exoskeleton. The Lokomat® FreeD (Hocoma AG, Switzerland) is an exoskeleton-type robot. Unlike the conventional Lokomat, the FreeD module allows pelvic translation to the right and left, along with rotation. These coordinated pelvic movements are mechanically facilitated by the device during walking. It is known that these movements are crucial for human walking and balance, and with the FreeD module, these pelvic movements have become part of robot-assisted gait training.

In a systematic review comparing Lokomat with conventional physiotherapy, it was reported that Lokomat is equally effective in terms of balance. Another review found that patients undergoing robot-assisted gait training showed better improvement in balance compared to those not receiving this treatment. The literature supports Lokomat's positive effects on both balance and walking.

In this research, virtual reality applications on Lokomat® will be integrated as part of the exercises in the Lokomat group and virtual reality-based balance training using the Balance Trainer will be employed for the Balance-Trainer group.

Patients will be allocated to the Lokomat and Balance-Trainer groups based on the treatment they receive. Both systems are actively used in the hospital, which research conduct, for the purpose of actively treating patients who meet the research criteria for improving balance and walking in stroke survivors. Participants will engage in exercises with Lokomat® or Balance Trainer for three weeks, five sessions per week, each session lasting 30 minutes, totaling 15 sessions, in addition to their current rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. Having the ICD-10 diagnosis code G.81 Hemiplegia
2. At least 3 weeks having passed since the diagnosis (Subacute and cronic periods)
3. Being 18 years of age or older
4. Having a Berg Balance Score between 21-40 (indicating an acceptable balance)
5. Being able to walk with or without support (FAC score of 2 or higher)

Exclusion Criteria:

1. Having a known additional neurological or orthopedic problem that could affect balance
2. Inability to adapt to virtual reality applications in Lokomat and Balance Trainer
3. Diagnosis being more than 2 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline and After last treatment seasion
  This is a simple and safe balance test designed to measure an individual's ability to maintain balance while performing functional tasks. The person is asked to perform 14 tasks, and scores are given based on the completion of each task. A score of 0 is assigned when the activity is not performed at all, while a score of 4 is given when the activity is completed independently. The highest possible score is 56, with 0-20 indicating balance impairment, 21-40 suggesting an acceptable balance, and 41-56 indicating good balance.
Spatiotemporal Gait Analysis | Baseline and After last treatment seasion
  In our research, spatiotemporal gait analysis will be conducted using the CMill VR+ device. As a result of gait analysis, parameters such as step lengths, swing, stance and double support phases, cadence, and levels of weight shifting to each side during walking will be recorded.

SECONDARY OUTCOMES:
Functional Independence Measure | Baseline and After last treatment seasion
  The Functional Independence Measure is a valid and reliable scale for assessing stroke patients, comprising 18 items that evaluate the patient both physically and cognitively. These items are primarily grouped under the headings of Self-Care, Sphincter Control, Transfer, Locomotion, Communication, and Social Cognition.
Functional Ambulation Category | Baseline and After last treatment seasion
  It assesses the amount of physical support needed during walking, scoring from 0 to 5, with observations made through the assessment. The scoring is based on the amount of support the patient requires, ranging from 0 - indicating inability to ambulate independently and requiring maximum support, to 5 - defining a patient who can walk independently on all surfaces.

OTHER OUTCOMES:
Patient Satisfaction | After last treatment seasion
  In the research, patient satisfaction was assessed using a scale ranging from 1 to 10. A higher score indicates better patient satisfaction. A score of 1 signifies complete dissatisfaction, while a score of 10 represents the highest level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided